CLINICAL TRIAL: NCT00416793
Title: A Phase II Study of Bortezomib in Combination With Carboplatin in Patients With Metastatic Pancreatic Cancer
Brief Title: Bortezomib and Carboplatin in Treating Patients With Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02894; NCI-2012-02894 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000522739; NO1-CM-17003-74; MDA-2006-0079 (Other: MD Anderson Cancer Network); 7752 (Other: CTEP); NCT00409877 (obsolete NCT alias)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bortezomib; Carboplatin

ARMS (1):
- Treatment (Experimental): Patients receive bortezomib IV on days 1, 4, 8, and 11 and carboplatin IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: carboplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
Drug: carboplatin — Given IV
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving bortezomib together with carboplatin works in treating patients with metastatic pancreatic cancer. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with carboplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate overall survival (OS) at 6 months with the combination of bortezomib and carboplatin in patients who previously received 1 prior regimen for metastatic pancreatic cancer.

SECONDARY OBJECTIVES:

I. To evaluate the objective tumor response rate, the duration of response, time to tumor progression, and overall survival.

II. To evaluate biological effects on peripheral blood mononuclear cells. III. To evaluate the safety profile of this combination. IV. To evaluate archival tissue for epithelial-to-mesenchymal transition (EMT) and E-cadherin and Zeb-1.

OUTLINE:

Patients receive bortezomib intravenously (IV) on days 1, 4, 8, and 11 and carboplatin intravenously (IV) over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma or carcinoma of the pancreas that is metastatic and not amenable to resection with curative intent
* Patients must have measurable disease defined by RECIST criteria; for the purpose of this study, primary mass in the pancreas is not considered as measurable disease
* Patients must have received one (1), and only one, prior systemic regimen for metastatic disease; patients who have received prior cisplatin or oxaliplatin are eligible; a systemic regimen administered for unresectable locally advanced disease that subsequently progressed to metastatic will be counted as 1 prior regimen; chemotherapy administered as adjuvant therapy or as a radiation sensitizer is not counted as a prior regimen
* Prior radiation is permitted; however, at least 3 weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all associated toxicities to NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 ≤ Grade 1 at the time of registration; measurable disease must be outside the previous radiation field or a new lesion inside the port must be present
* At least two weeks must have elapsed since any major surgery and patients must have recovered from all associated toxicities to ≤ CTCAE Grade 1 at the time of registration
* At least 4 weeks must have elapsed since previous chemotherapy except for regimens that are administered on a daily, weekly, or every other week schedule, in which case at least 2 weeks must have elapsed since previous chemotherapy; patients must have recovered from all associated toxicities to CTCAE ≤ Grade 1 at the time of registration
* ECOG performance status =< 1 (Karnofsky >= 70%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin ≥ 9 g/dl
* Total bilirubin =<1.5 X institutional upper limit of normal
* AST (SGOT) & ALT (SGPT) =< 2.5 X institutional upper limit of normal or =< 5 X institutional upper limit of normal if patient has liver metastasis
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance >= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Other prior malignancy is allowed as long as the patient does not require active treatment for their second malignancy and there is no radiographic evidence of second malignancy; patients who are receiving hormonal therapy for breast or prostate cancer as adjuvant treatment are eligible
* The effects of bortezomib on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because carboplatin, the other therapeutic agent used in this trial, is known to be teratogenic, women of child-bearing potential and men of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document; written informed consent must be obtained prior to any evaluations being performed solely for the purposes of screening for eligibility for this study

Exclusion Criteria:

* Patients who have only locally advanced disease (not metastatic) are excluded
* Patients who have received prior treatment with carboplatin, bortezomib, or another proteasome inhibitor are excluded
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; however, brain imaging studies are not required to assess eligibility if the patient has no neurological signs or symptoms
* Patients with current neurotoxicity, defined as greater than CTCAE Grade 1 neurotoxicity
* Patients must not be planning to receive any other concomitant anticancer treatment including chemotherapy, radiation therapy, biologic agents, or any other investigational drugs
* Patients must not have significant history of cardiac disease, i.e., unstable angina, congestive heart failure with New York Heart Association class 3 or 4, and myocardial infarction within the last 6 months
* Pregnant women are excluded from this study because bortezomib is a proteasome inhibitor agent with the potential for teratogenic or abortifacient effects; carboplatin has been shown to be embryotoxic and teratogenic in rats; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bortezomib and carboplatin, breastfeeding should be discontinued if the mother is treated with these drugs
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with bortezomib and carboplatin; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gauri Varadhachary, Principal Investigator — MD Anderson Cancer Network
Locations (1):
- MD Anderson Cancer Network, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: December 7, 2006 to August 26, 2008. All recruitment was done at UT MD Anderson Cancer Center.
Pre-assignment Details: The study was terminated early since the protocol met prospective criteria for early stopping.
Groups:
- Bortezomib + Carboplatin: Bortezomib 1.3 mg/m2 by vein (IV) on days 1, 4, 8 + 11; Carboplatin Area Under the Curve (AUC) of 5 IV over 30 minutes
Period: Overall Study
Arm/Group | Bortezomib + Carboplatin
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib + Carboplatin
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 49 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 6 Months
Description: Overall survival (OS) at 6 months with the combination of bortezomib and carboplatin in participants who previously received 1 prior regimen for metastatic pancreatic cancer from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months. Rate equals number of participants living at 6 months following treatment divided by the total number of participants.
Time Frame: up to 6 months
Population: Analysis was per protocol; Limited analysis due to study early termination.
Measure: Number; unit: Proportion of participants
Arm/Group | Bortezomib + Carboplatin
Number analyzed (Participants) | 9
Proportion of participants | 0

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate measured by number of patients per the total treatment population who partially or completely responded to treatment. Participants reevaluated for response every 6 weeks. In addition to a baseline scan, confirmatory scans at 4 weeks following initial documentation of objective response.
Time Frame: from assignment of treatment until the date of first documented progression, assessed up to 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib + Carboplatin
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: 17 months
Arm/Group | Bortezomib + Carboplatin
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Carboplatin (N=9)
Abdominal Pain (Gastrointestinal disorders) | 4
Alopecia (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Aspartate Aminotransferase increased (Metabolism and nutrition disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Bilirubin increased (Metabolism and nutrition disorders) | 1
Blood Glucose Increase (Metabolism and nutrition disorders) | 4
Blood uric acid increased (Metabolism and nutrition disorders) | 1
Blurred vision (Eye disorders) | 1
Cardiac Pain (Cardiac disorders) | 2
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Creatinine increased (Metabolism and nutrition disorders) | 1
Depression (Nervous system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Erythema multiform (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 5
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Headache (General disorders) | 1
Increased Alkaline Phosphatase (Metabolism and nutrition disorders) | 5
Insomnia (General disorders) | 2
Mucositis (oral) (Gastrointestinal disorders) | 1
Myocardial Ischemia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Pain(back) (Musculoskeletal and connective tissue disorders) | 2
Peripheral Sensory Neuropathy (Musculoskeletal and connective tissue disorders) | 2
Plate Count decrease (Blood and lymphatic system disorders) | 5
Renal(loss of feeling of urination) (Renal and urinary disorders) | 1
Serum Sodium increased (Metabolism and nutrition disorders) | 1
Serum magnesium decreased (Metabolism and nutrition disorders) | 1
Taste Alteration (General disorders) | 4
Thrombosis (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 4

LIMITATIONS AND CAVEATS:
Given the toxicity and lack of objective responses observed with this regimen, the protocol met prospective criteria for early stopping and was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less